CLINICAL TRIAL: NCT02263391
Title: Collaborative Biosocial Research on HIV Risk and Prevention in Women
Brief Title: HIV Risk and Prevention in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Russian Foundation for Basic Research (RFBR) (Unknown); Saint Petersburg State University, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3878; 1R21AA022596-01 (NIH)
Record Dates: First submitted 2014-09-26; First posted 2014-10-13 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: HIV
Keywords: transmission; prevention; women; childbearing age; HIV testing; testing strategy
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Opt-in testing (Experimental): Common barriers to HIV screening testing will be removed as much as possible (i.e., providing rapid testing, results shortly available, testing on-site, confidentiality). The research assistant will say: "There is voluntary HIV testing available to all study participants if you wish to do it. It is free, private, it is only a finger stick, and you will learn your HIV results in just minutes." Participants will be scheduled for a two-hour appointment to complete the written consent procedure, enroll in the study, and participate in the study activities, testing and a focus group.
  Interventions: Behavioral: Opt-in or Opt-out testing; Behavioral: Focus Group
- Opt-out testing (Experimental): Participants will be informed that a routine health test bundle is available on a voluntary basis to study participants, and the participant may elect to decline all or any individual part of the testing. The assistant will say: "We are offering a voluntary panel of routine health screening test today for study participants. It includes blood sugar, cholesterol, and HIV. We recommend all of them for everyone, but you can choose to decline any or all of them. This is free, private, it is only a finger stick, and you will learn your results for all the tests in just minutes." Participants will be scheduled for a two-hour appointment to complete the written consent procedure, enroll in the study, and participate in the study activities, testing and a focus group.
  Interventions: Behavioral: Opt-in or Opt-out testing; Behavioral: Focus Group

INTERVENTIONS:
Behavioral: Opt-in or Opt-out testing — Study participants will be offered a health screening onsite.
Behavioral: Focus Group — Study participants will be invited to participate in a focus group discussion.

SUMMARY:
This study gathers information about HIV testing utilization and influences on HIV testing decisions among young, general population Russian women at-risk of HIV exposure. The study compares HIV testing acceptance across two types of low-barrier testing strategies (opt-in vs. opt-out) and conducts one of the first randomized experimental comparisons of these strategies. The overarching goal is to gain knowledge that can be used to increase utilization of HIV testing among at-risk young women and offer gender-specific strategies for improving prevention.

DETAILED DESCRIPTION:
The study uses an adaptive design. That is, the procedures and phases of the study experienced by a participant depend to some extent on their responses to earlier phases. Ultimately, this design yields a number of practice relevant pathways and endpoints, each of which has a testing rate associated with it.

Phase-I is initial screening for risk status, collecting background data, and ascertaining whether there has been recent independent HIV testing. If there has been independent testing, information about the independent testing is collected and the participant's involvement is complete.

Those who are not independent testers enter Phase-II. Phase II will include: randomization to opt-in vs. opt-out conditions; a survey asking about reasons for acceptance or non-acceptance; participating in a focus group in which participants who have not accepted HIV testing (non-accepters) and those who accepted (accepters) will be asked to discuss their health beliefs related to HIV prevention, barriers and reasons for testing/not testing; then (5) after the focus group is complete, privately offer another testing opportunity to non-accepters, under the same opt-in or opt-out strategy to which they previously were randomized. The design was selected in order simultaneously answer a number of questions that we believe will be important for engineering a testing and prevention strategy suitable for testing in a subsequent study: (1) identify key attitudes, beliefs and knowledge (survey); (2) contrast opt-in and opt-out strategies (randomized trial); (3) generate qualitative data about reasons for decisions in the women's own words (focus group); and (4) identify any incremental benefit related to peer discussion.

ELIGIBILITY:
Inclusion Criteria:

* The participant's sexual risk behaviors (i.e., a) two or more partners in the last 12 months, or her partner's HIV risk (e.g., HIV positive, no HIV testing and a diagnosis of sexually transmitted diseases in last 12 months, multiple partners, blood transmission, male partners, served in prison, or drug use) and no or inconsistent condom use in the last 3 months, and no HIV testing in the last 12 months, or b) any sexually-transmitted disease and no HIV testing in the last 12 months).

Exclusion Criteria:

* Does not speak Russian, are currently pregnant, have a condition that might preclude a finger-stick procedure, or have tested HIV positive in the past.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who accepted a rapid health screening/HIV test | At first visit, an expected average of 1 hour
  Women's decision to take/not take a health screening test/HIV test is recorded. If a woman chooses to be tested, she will be asked a few questions to assess her reasons for being tested. She will be provided with the results of the testing. If a woman's test is positive for HIV (or other health risks in the bundled opt-out condition), counseling with a trained study nurse, physician or psychologist will be available on-site and a referral for additional testing, counseling, and appropriate medical care will be provided.
Number of participants who accepted the health screening/HIV test after a focus group | After completing a focus group discussion, an expected average of 4 weeks
  participating in a focus group in which participants who have not accepted HIV testing (non-accepters) and those who accepted (accepters) will be asked to discuss their health beliefs related to HIV prevention, barriers and reasons for testing/not testing; then (5) after the focus group is complete, privately offer another testing opportunity to non-accepters, under the same opt-in or opt-out strategy to which they previously were randomized.

SECONDARY OUTCOMES:
Brief survey to assess reasons for being tested | At first visit, an expected average of 1 hour
  Participants who accepted a rapid health screening/HIV test are asked about reasons for taking the test at this time.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Balachova, PhD, Principal Investigator — University of Oklahoma; Alla Shaboltas, PhD, Principal Investigator — Facility: St. Petersburg State University St. Peterburg, Russian Federation
Locations (2):
- University of Oklahoma, Oklahoma City, Oklahoma, United States
- St. Petersburg State University, Saint Peterburg, Russia

REFERENCES:
- [Background] Balachova TN, Batluk JV, Bryant KJ, Shaboltas AV. International collaboration in HIV prevention research: evidence from a research seminar in Russia. AIDS Res Hum Retroviruses. 2015 Feb;31(2):163-72. doi: 10.1089/AID.2014.0078. Epub 2014 Dec 31. PMID 25430518